CLINICAL TRIAL: NCT03554798
Title: A Phase 2 Study to Evaluate the Safety and Immunogenicity of Two Novel Oral Polio Type 2 (nOPV2) Vaccine Candidates in Healthy Children Aged 1 to 5 Years and in Healthy Bivalent Oral Polio Vaccine-inactivated Polio Vaccine (bOPV-IPV) Vaccinated Infants
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Novel Oral Polio Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M5 ABMG
Record Dates: First submitted 2018-05-08; First posted 2018-06-13 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Allocation of each subject to a given group will be described in a computer-generated randomization schedule. Based on this randomization code, the study vaccine will be packaged and labeled. Medication code numbers will be preprinted on the study vaccine labels and assigned as subjects qualify for the study and are randomly assigned to dosing schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nOPV2 Candidate 1 (monovalent oral poliovirus type1) (Experimental): Cohort A: IPV and/or OPV vaccinated participants aged 1 to 5 years vaccinated with candidate 1.
  Cohort B: 6 weeks Infants vaccinated with 3 doses of bOPV and 1 dose of IPV, followed with 1 dose of candidate 1.
  Interventions: Biological: nOPV2 (monovalent oral polio vaccine)
- nOPV2 Candidate 2 (monovalent oral poliovirus type2) (Experimental): Cohort A: IPV and/or OPV vaccinated participants aged 1 to 5 years vaccinated with candidate 2.
  Cohort B: Infants vaccinated with 3 doses of bOPV and 1 dose of IPV, followed with 1 dose of candidate 2.
  Interventions: Biological: nOPV2 (monovalent oral polio vaccine)

INTERVENTIONS:
Biological: nOPV2 (monovalent oral polio vaccine) — Cohort A: 150 IPV and/or OPV vaccinated participants aged 1 to 5 years vaccinated with candidate 1 or 2; two 10‸6 CCID50 (50% cell culture infective dose) doses separated by 28 days.
  Cohort B: 972 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 10‸5 CCID50 dose of candidate 1 or 2.

SUMMARY:
This will be a single center, age de-escalation, partly-blinded, randomized study.

The trial will be performed with the participation of 100 healthy children age 1-5 years who have been vaccinated with inactivated polio vaccine (IPV) and/or oral polio vaccine (OPV) in their first year of life and of 648 healthy 6 week-old infants, who will be pre-vaccinated with bOPV-IPV before being randomized to study groups. The allocation of 18-22 week-old infants to groups will be performed in a randomized manner. Following completion and Data Safety Monitoring Board (DSMB) review of follow-up for general safety data (Serioius Adverse Events -SAEs-, Important Medical Events -IMEs- and severe adverse events -AEs), a DSMB recommendation to proceed will result in randomization of the final cohort of infants. Allocation of 1 to 5 year-old children to groups will be performed in a randomized manner.

The DSMB will establish and continuously assess stopping rules for safety.

ELIGIBILITY:
Inclusion Criteria:

1. For Cohort A children enrolled at 1 to 5 years of age who have previously been fully vaccinated according to MoH recommendations with OPV and/or IPV.
2. For Cohort B infants enrolled at 6 weeks of age (-1, + 2 weeks) with birth weight >2,500 gm. To be eligible to continue into the experimental phase of the study infants must be vaccinated with 3 doses of bOPV and one dose of IPV prior to administration of the study vaccine at 18-22 weeks of age to take into account the visit windows for enrollment (age 6 weeks, -1 or + 2 weeks) and subsequent OPV vaccination windows (± 1 week). The last polio vaccine must have been administered at least 4 weeks prior to the first dose of study vaccine. Subjects in Cohort B who do not complete the three routine vaccination visits will be replaced in the study, and their parents/guardians will be encouraged to complete the primary vaccinations series.
3. Healthy children without obvious medical conditions like immunodeficiency diseases, severe congenital malformations, severe neurological diseases or any other disease that require high doses of corticosteroids or immunotherapies that preclude the subject to be in the study as established by the medical history and physical examination.
4. Written informed consent obtained from 1 or 2 parent(s) or legal guardian(s) as per country regulations.

Exclusion Criteria:

1. For all participants the presence of anyone under 10 years of age in the subject's household (living in the same house or apartment unit) who does not have complete "age appropriate" vaccination status with respect to poliovirus vaccines at the time of study vaccine administration. For household members younger than 18 months age appropriate vaccination is at least three (3) doses of IPV. For household members between 18 months and 10 years "age appropriate" vaccination is at least three (3) doses of IPV or tOPV plus one (1) booster dose of any antipolio vaccine.
2. For all participants having a member of the subject's household (living in the same house or apartment unit) who is under 6 months of age at the moment of study vaccine administration.
3. For all participants having a member of the subject's household (living in the same house or apartment unit) who has received OPV in the previous 3 months before study vaccine administration.
4. For Cohort A: receipt of polio vaccines within the 3 months prior to the administration of the study vaccine (number of previous polio vaccine doses to be documented). Any other vaccine 4 weeks before study entry.
5. For Cohort A: any participating children attending day care or pre-school during their participation in the study until one month after their last nOPV2 administration.
6. For Cohort B: any receipt of polio vaccines prior to administration of the study vaccine other than 3 doses of bOPV and 1 dose of IPV.
7. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus (HIV) infection in the potential participant or any member of the subject's household.
8. Family history of congenital or hereditary immunodeficiency.
9. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
10. Known allergy to any component of the study vaccines or to any antibiotics, that share molecular composition with the nOPV2 vaccines.
11. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections (of IPV).
12. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
13. Acute severe febrile illness at day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all inclusion criteria are met.).
14. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1025 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Panama (2):
  - Cevaxin Vaccination Center, David, Chiriquí Province
  - Cevaxin Vaccination Center, Panama City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wahid R, Mercer LD, De Leon T, DeAntonio R, Saez-Llorens X, Macadam A, Chumakov K, Strating J, Koel B, Konopka-Anstadt JL, Oberste MS, Burns CC, Andino R, Tritama E, Bandyopadhyay AS, Aguirre G, Ruttimann R, Gast C, Konz JO. Genetic and phenotypic stability of poliovirus shed from infants who received novel type 2 or Sabin type 2 oral poliovirus vaccines in Panama: an analysis of two clinical trials. Lancet Microbe. 2022 Dec;3(12):e912-e921. doi: 10.1016/S2666-5247(22)00254-3. Epub 2022 Nov 1. PMID 36332645
- [Derived] Saez-Llorens X, Bandyopadhyay AS, Gast C, Leon T, DeAntonio R, Jimeno J, Caballero MI, Aguirre G, Oberste MS, Weldon WC, Konopka-Anstadt JL, Modlin J, Bachtiar NS, Fix A, Konz J, Clemens R, Costa Clemens SA, Ruttimann R. Safety and immunogenicity of two novel type 2 oral poliovirus vaccine candidates compared with a monovalent type 2 oral poliovirus vaccine in children and infants: two clinical trials. Lancet. 2021 Jan 2;397(10268):27-38. doi: 10.1016/S0140-6736(20)32540-X. Epub 2020 Dec 9. PMID 33308427

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage I - Group A2H2: 50 polio vaccine primed children aged 1 to <5 years were to receive two 106 CCID50 doses of nOPV2 candidate 2, 2016, separated by 28 days (Group A2H2[2016]).
- Stage II - A1H2 [2018]: 50 IPV and/or OPV vaccinated participants aged 1 to 5 years administered with two 106 CCID50 doses of candidate 1 (2018) separated by 28 days.
- Stage II - A2H2 [2018]: 50 IPV and/or OPV vaccinated participants aged 1 to 5 years administered with two 106 CCID50 doses of candidate 2 (2018) separated by 28 days.
- Stage I -- Group B2L1+L2[2016]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 105 CCID50 dose of candidate 2 (2016). 50 randomly selected subjects from group B2L1 received a second 105 CCID50 dose of candidate 2 (2016), 28 days later.
- Stage I - B2H1+H2[2016]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 106 CCID50 dose of candidate 2 (2016).50 infants randomly selected from B2H1[2016] to receive a second 106 CCID50 dose of candidate 2 (2016), 28 days later.
- Stage II - Group B1L1+L2[2018]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) administered with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 105 CCID50 dose of candidate 1 (2018).
- Stage II - Group B1H1+H2[2018]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 106 CCID50 dose of candidate 1.50 infants randomly selected to receive a second 106 CCID50 dose of candidate 1, 28 days later
- Stage II - Group B2L1+L2 [2018]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 105 CCID50 dose of candidate 2 [2018].50 infants randomly selected to receive a second 105 CCID50 dose of candidate 2 [2018], 28 days later.
- Stage II - Group B2H1+H2[2018]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 106 CCID50 dose of candidate 2 [2018].50 infants randomly selected to receive a second 106 CCID50 dose of candidate 2 [2018], 28 days later.
Period: Overall Study
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1+L2 [2018] | Stage II - Group B2H1+H2[2018]
Started | 50 | 50 | 51 | 156 | 144 | 138 | 150 | 135 | 151
Completed | 45 | 47 | 48 | 154 | 141 | 137 | 149 | 133 | 149
Not Completed | 5 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Stage I -- Group B2L1+L2[2016]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 105 CCID50 dose of candidate 2 (2016).50 infants randomly selected from B2L1[2016] to receive a second 105 CCID50 dose of candidate 2 (2016), 28 days later.
- Stage II - Group B1L1+L2[2018]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) administered with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 105 CCID50 dose of candidate 1 (2018).50 infants randomly selected to receive a second 105 CCID50 dose of candidate 1 (2018), 28 days later
- Stage II - Group B2L1 +L2[2018]: 162 infants enrolled at 6 weeks of age (-7 to +14 days) vaccinated with 3 doses of bOPV at 6, 10 and 14 weeks of age and 1 dose of IPV at 14 weeks of age, followed at 18-22 weeks of age with one 105 CCID50 dose of candidate 2 [2018].50 infants randomly selected to receive a second 105 CCID50 dose of candidate 2 [2018], 28 days later.
- Total: Total of all reporting groups
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1 +L2[2018] | Stage II - Group B2H1+H2[2018] | Total
Number analyzed (Participants) | 50 | 49 | 51 | 156 | 144 | 138 | 150 | 135 | 151 | 1024
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 49 | 51 | 156 | 144 | 138 | 150 | 135 | 151 | 1024
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 29 | 66 | 65 | 69 | 71 | 74 | 73 | 488
  Male | 33 | 25 | 22 | 90 | 79 | 69 | 79 | 61 | 78 | 536
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mixed race | 24 | 49 | 51 | 151 | 141 | 135 | 147 | 132 | 151 | 981
  Other | 26 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26
  Black or African American | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 5
  Central American Indian | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 1 | 0 | 9
  Hispanic | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Panama | 50 | 49 | 51 | 156 | 144 | 138 | 150 | 135 | 151 | 1024

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Reactions (SARs), Severe AEs and Important Medical Reactions (IMRs) Incidence
Description: Number of subjects experiencing Serious Adverse Reactions (SAR), severe AR and IMR, i.e. SAEs, severe AEs (grade 3), or IMEs considered consistent with a causal association with study vaccines as of the informed consent signature date and throughout the study period in all groups.
Time Frame: 6 months
Population: Safety parameters were tabulated and analyzed descriptively in the total vaccinated (TV) population, according to the actual vaccine received. TV population is defined as all subjects who received at least one dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1 +L2[2018] | Stage II - Group B2H1+H2[2018]
Number analyzed (Participants) | 50 | 49 | 51 | 155 | 144 | 138 | 150 | 135 | 151
participants | 0 | 1 | 0 | 5 | 6 | 1 | 1 | 1 | 1

2. Primary Outcome: Single Dose Seroprotection Rate
Description: Seroprotection rate of type 2 polio neutralizing antibodies at Day 28 following a single 105 or 106 CCID50 dose of nOPV2 candidates in all groups. Seroprotection rate is defined as the percentage of subjects with type 2-specific antibody titers ≥ 1:8 per group.
Time Frame: 2 months
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1+L2 [2018] | Stage II - Group B2H1+H2[2018]
Number analyzed (Participants) | 45 | 37 | 47 | 145 | 136 | 131 | 143 | 127 | 146
Participants | 45 | 37 | 47 | 125 | 132 | 122 | 134 | 115 | 138

3. Secondary Outcome: Any Other SAEs, AEs and IMEs Incidence
Description: Number of participants experiencing any other SAE, any solicited AE, any unsolicited AEs and any IME as well as any clinical laboratory deviation considered consistent with causal association to study vaccine (primary objective) following one or two doses of either nOPV2 candidates.
Time Frame: 6 months
Population: Assessed in total vaccinated (TV) population, defined as all subjects who received at least one dose of study vaccine.Only secondary objectives included intent to compare the M5 data with the control sample which had received Sabin mOPV2 in M2 study (NCT02521974-historical control for M5).
  Extent of exposure: in M5 Stage II, the second dose of study vaccine were received by 47 (94%) children in Group A1H2[2018] and 50 (98%) children in Group A2H2[2018].
Measure: Number; unit: participants
Groups:
- M2 Group 2+3: 114 infants (3 bOPV/1 IPV primed) were to receive at 18 weeks of age one dose of Sabin mOPV2 (at a titer of ≥ 105 CCID50) (Group 2). A randomly selected sub-group of 50 infants were to receive a second dose of Sabin mOPV2 approximately 28 days later (Group 3).
- M2 Children: 50 IPV and/or OPV vaccinated children aged 1 to <5 years were to receive 2 doses of Sabin mOPV2 (at a titer of ≥ 105 CCID50) (Group 1), separated by 28 days
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1+L2 [2018] | Stage II - Group B2H1+H2[2018] | M2 Group 2+3 | M2 Children
Number analyzed (Participants) | 50 | 49 | 51 | 155 | 144 | 138 | 150 | 135 | 151 | 110 | 50
participants
  SAEs | 0 | 1 | 2 | 2 | 0 | 9 | 1 | 3 | 5 | 0 | 1
  IMEs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AEs | 32 | 36 | 44 | 30 | 29 | 34 | 37 | 36 | 33 | 36 | 28

4. Secondary Outcome: Seroconversion Rates Comparison
Description: Seroconversion rates against type 2 of one or two 106 CCID50 doses of both nOPV2 vaccine candidates in healthy children aged 1 to 5 years and of two doses of both nOPV2 vaccine candidates at both 105 and 106 CCID50 dose levels at approximately 22 weeks of age in infants previously vaccinated with 3 doses of bOPV and 1 dose of IPV, and compare this immunogenicity with a control sample of participants receiving the same vaccination schedule followed by one or two doses of Sabin mOPV2 in a prior study (M2) designed and performed to serve as a control for the current study. Seroconversion is defined as a change from seronegative to seropositive, and in seropositive subjects, as an antibody titer increase of ≥ 4 fold over baseline (Day 0) titers corrected for maternal antibodies titers where applicable/age-appropriate.
Time Frame: 2 months
Population: Subset of subjects with baseline immunity (NAb titer) sufficiently low to enable observation of seroconversion (≤8.5 log2 i.e. ≤4-fold from assay ULOQ) at D56. Only secondary objectives included intent to compare the M5 data with the control sample of similarly aged infants and young children who had received Sabin mOPV2 in a M2 study, which was designed to serve as a historical control for M5.
  For further details on results corresponding to M2 study, please refer to NCT02521974.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1+L2 [2018] | Stage II - Group B2H1+H2[2018] | M2 Group 2+3 | M2 Children
Number analyzed (Participants) | 19 | 17 | 23 | 42 | 45 | 45 | 48 | 44 | 48 | 39 | 9
Participants | 18 | 17 | 22 | 40 | 43 | 44 | 47 | 38 | 48 | 38 | 6

5. Secondary Outcome: Seroprotection Rates Comparison
Description: Seroprotection rates against type 2 of one or two 106 CCID50 doses of both nOPV2 vaccine candidates in healthy children aged 1 to 5 years and of two doses of both nOPV2 vaccine candidates at both 105 and 106 CCID50 dose levels at approximately 22 weeks of age in infants previously vaccinated with 3 doses of bOPV and 1 dose of IPV, and compare this immunogenicity with a control sample of participants receiving the same vaccination schedule followed by one or two doses of Sabin mOPV2 in a prior study (M2) designed and performed to serve as a control for the current study.
  Seroprotection rate is defined as the percentage of subjects with type 2-specific neutralizing antibody titers ≥ 1:8 per group.
Time Frame: 2 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1+L2 [2018] | Stage II - Group B2H1+H2[2018] | M2 Group 2+3 | M2 Children
Number analyzed (Participants) | 44 | 39 | 46 | 44 | 47 | 46 | 48 | 44 | 48 | 40 | 46
Participants | 44 | 39 | 46 | 44 | 46 | 45 | 48 | 43 | 48 | 39 | 46

6. Secondary Outcome: Viral Shedding
Description: Level of viral shedding in stool at fixed time points following administration of one or two doses of both nOPV2 candidates at both 105 and 106 CCID50 dose levels in infants at approximately 18-22 weeks of age after having been previously vaccinated with 3 doses of bOPV and 1 dose of IPV, and compare this shedding to a control sample of participants receiving the same vaccination schedule followed by one or two doses of Sabin mOPV2 in a prior study designed to serve as a control for the current study.
  This is determined by measuring the median number of days taken to get stool cultures negative for poliovirus presence (TTCN stands for median time to culture negative). Kaplan-Meier methods were used to describe the time to cessation of shedding for any shedding (PCR detection).
Time Frame: 2 months
Population: Subset of subjects corresponding to 2018 Candidates cohorts. 2016 Candidate cohorts did not participate on this endpoint assessment.
  Only secondary objectives included intent to compare the M5 data with the control sample of similarly aged infants and young children who had received Sabin mOPV2 in a M2 study, which was designed to serve as a historical control for M5.
  For further details on results corresponding to M2 study, please refer to NCT02521974.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1+L2 [2018] | Stage II - Group B2H1+H2[2018] | M2 Group 2+3 | M2 Children
Number analyzed (Participants) | 0 | 46 | 51 | 0 | 0 | 125 | 140 | 124 | 141 | 91 | 48
days |  | 5 [4 to 5] | 3 [2.5 to 5] |  |  | 6 [5 to 7] | 6 [5 to 7] | 6 [5 to 7] | 5 [4 to 6] | 6 [5 to 7] | 6.5 [5 to 9]

7. Secondary Outcome: Neurovirulence
Description: Potential for neurovirulence of virus isolated from a subset of stool samples of infants at approximately 18-22 weeks of age after having been previously vaccinated with 3 doses of bOPV and 1 dose of IPV, and following a single dose of both nOPV2 candidates at the 106 CCID50 dose level, as measured in an animal model, and compare this with a control sample (M2 study).
  For each of the children / infants receiving a 106 CCID50 dose of the 2018 cohorts as well as all participants in study M2, an exploratory endpoint sample (EES) of poliovirus shed in stools following the first dose was identified, if possible, with which to perform a modified neurovirulence test in a transgenic mouse model. Data from each sample tested was summarized by group per vaccine candidate. The proportion of mice paralyzed and the odds ratio of paralysis from the single-dose assay were the primary means of comparison of neurovirulence of shed virus between each candidate and the Sabin mOPV2 control samples.
Time Frame: 2 months
Population: Per the description under the Outcome Measure Description section, these groups do not match the participants arms distribution, as these results are related to the vaccine candidates behaviour in mice, not to the participating subjects.
  Only secondary objectives included intent to compare the M5 data with the control sample of M2 study, which was designed to serve as a historical control for M5. For further details on results corresponding to M2 study, please refer to NCT02521974.
Measure: Number; unit: percentage of neurovirulence
Units Other Than Participants: EES
Groups:
- mOPV2: Monovalent Oral Polio Vaccine
- nOPV2 C1 2018; nOPV2 C2 2018: Novel Oral Polio Vaccine Candidate 1 - 2018
Arm/Group | mOPV2 | nOPV2 C1 2018 | nOPV2 C2 2018
Number analyzed (Participants) | 5 | 22 | 29
Number analyzed (EES) | 5 | 22 | 29
percentage of neurovirulence | 90 | 0 | 30

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Stage I - Group A2H2 | Stage II - A1H2 [2018] | Stage II - A2H2 [2018] | Stage I -- Group B2L1+L2[2016] | Stage I - B2H1+H2[2016] | Stage II - Group B1L1+L2[2018] | Stage II - Group B1H1+H2[2018] | Stage II - Group B2L1+L2 [2018] | Stage II - Group B2H1+H2[2018]
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 0/51 | 0/155 | 0/144 | 0/138 | 0/150 | 0/135 | 1/151
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/49 | 3/51 | 7/155 | 1/144 | 14/138 | 14/150 | 9/135 | 15/151
Other Adverse Events (participants affected / at risk) | 40/50 | 36/49 | 44/51 | 82/155 | 93/144 | 129/138 | 127/150 | 118/135 | 126/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage I - Group A2H2 (N=50) | Stage II - A1H2 [2018] (N=49) | Stage II - A2H2 [2018] (N=51) | Stage I -- Group B2L1+L2[2016] (N=155) | Stage I - B2H1+H2[2016] (N=144) | Stage II - Group B1L1+L2[2018] (N=138) | Stage II - Group B1H1+H2[2018] (N=150) | Stage II - Group B2L1+L2 [2018] (N=135) | Stage II - Group B2H1+H2[2018] (N=151)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 9 | 8 | 2 | 10
Soft Tissue Abscess (preauricular) (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0
Urticaria (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 1 | 4 (7) | 6 | 4 | 3
Second degree burn (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonic clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Acute Diarrheal Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular Septal Defect (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Withlow left hand (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Congeniital Cortical Blindness (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage I - Group A2H2 (N=50) | Stage II - A1H2 [2018] (N=49) | Stage II - A2H2 [2018] (N=51) | Stage I -- Group B2L1+L2[2016] (N=155) | Stage I - B2H1+H2[2016] (N=144) | Stage II - Group B1L1+L2[2018] (N=138) | Stage II - Group B1H1+H2[2018] (N=150) | Stage II - Group B2L1+L2 [2018] (N=135) | Stage II - Group B2H1+H2[2018] (N=151)
Irritability (General disorders) | 2 | 3 | 5 | 30 | 18 | 23 | 27 | 25 | 25 — Solicited AE
Abnormal crying (General disorders) | 2 | 7 | 5 | 35 | 24 | 26 | 24 | 21 | 25 — Solicited AE
Fever (General disorders) | 6 | 12 | 15 | 14 | 12 | 15 | 12 | 20 | 18 — Solicited AE
Loss of Appetite (General disorders) | 16 | 13 | 13 | 22 | 13 | 11 | 15 | 14 | 19 — Solicited AE
Vomiting (Gastrointestinal disorders) | 6 | 5 | 6 | 20 | 21 | 19 | 22 | 20 | 19 — Solicited AE
Drowsiness (General disorders) | 2 | 9 | 5 | 8 | 9 | 6 | 11 | 10 | 15 — Solicited AE
Influenza (Infections and infestations) | 9 | 23 | 25 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 4 | 7 | 8 | 1 | 1 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 9 | 4 | 9 | 7 | 2 | 9 | 1 | 4
Nasopharyngitis (Infections and infestations) | 18 | 2 | 4 | 52 | 65 | 62 | 71 | 69 | 78
Gastroenteritis (Infections and infestations) | 2 | 6 | 6 | 1 | 2 | 4 | 2 | 2 | 1
Rhinitis (Infections and infestations) | 5 | 5 | 5 | 11 | 8 | 5 | 3 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Otitis (Infections and infestations) | 0 | 3 | 4 | 0 | 3 | 1 | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 4 | 6 | 3 | 2 | 1 | 6
Bronchitis (Infections and infestations) | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Varicella (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Teething (Gastrointestinal disorders) | 1 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 1 | 7 | 1 | 9
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 0 | 1 | 3 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 4 | 7 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 2 | 4 | 1 | 4
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 2 | 0
Viral Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 9 | 3 | 0 | 1 | 0 | 5
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 4 | 5 | 5 | 6
Normocytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 2 | 6 | 10 | 5 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 5 | 5
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 0
Infantile Colic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Overweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2 | 2 | 3 | 7 | 4
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Milk Allergy (Immune system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Transaminases increase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gross Motor Delay (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurodevelopmental Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
External Ear Inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess Jaw (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amoebiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amoebic Dysentery (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Roseola (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Spinal Cord Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Psychomotor Retardation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Motor Developmental Delay (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blindness Cortical (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected Bite Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03554798/Prot_SAP_000.pdf